CLINICAL TRIAL: NCT06675552
Title: PHenotype-based RApid SEquencing of Guideline-directed Medical Therapy for Heart Failure With Reduced Ejection Fraction (PHRASE-HF): A Multicentre, Prospective, Non-interventional Study to Examine Outcomes of Rapid In-hospital Implementation of GDMT and Its Translation From Discharge Into Routine Care
Brief Title: Non-interventional Study on Guideline Directed Medical Therapy for Patients With Heart Failure (HF) in Germany
Acronym: PHRASE-HF
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D1699R00045
Record Dates: First submitted 2024-09-20; First posted 2024-11-05 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Heart Disease; Heart Failure; Cardiovascular Disease; Heart Failure, Systolic
Keywords: Heart Failure with Reduced Ejection Fraction (HFrEF); Guideline Directed Medical Therapy; Real-World Evidence
MeSH Terms: conditions — Heart Diseases; Heart Failure; Cardiovascular Diseases; Heart Failure, Systolic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Heart failure (HF) is a global public health issue that affects more than 63 million people worldwide. The clinical and economic burden of HF on health care systems is substantial. Heart failure with reduced ejection fraction (HFrEF) represents approximately 50% of the HF patient population.The burden of HF is expected to increase substantially as the population ages, and despite improvements in treatment, hospitalisation and mortality rates remain especially high in HFrEF patients. The current guideline recommendation of directed medical therapy for HFrEF combines four drug classes with proven prognostic benefit: Angiotensin receptor-neprilysin inhibitor (ARNI)/angiotensin converting enzyme inhibitors (ACE I)/angiotensin receptor blockers (ARB), betablockers (BB), mineralocorticoid receptor antagonists (MRA), and sodium-glucose co-transporter 2 inhibitors (SGLT2i). The 2023 ESC (European Society of Cardiology) HF guideline update additionally recommends a rapid in-hospital sequencing approach of guideline-directed medical therapy (GDMT) with frequent physician visits during the first 6 weeks post discharge. Studies investigating the implementation of GDMT in a real-world setting have shown that a significant proportion of patients did not receive the recommended drug combination therapy. Delayed initiation of GDMT contributes to the low number of patients receiving guideline concordant HFrEF therapy, which ultimately may affect patient outcomes. One approach to implement the 2023 ESC guideline updates for heart failure treatment regarding early in-hospital initiation and rapid up-titration of GDMT could be to provide specific training on GDMT recommendations. Such a standardised training is offered to the physicians treating HF patients within selected hospitals of the German Helios hospital network (Helios-GDMT-program). Evidence is needed in order to assess whether in-hospital initiation and up-titration of all phenotype concordant classes of GDMT at hospital discharge can be observed after standardised physician training and whether the GDMT-program implementation also translates into real-world routine outpatient care with respect to use of GDMT and clinical outcomes.

DETAILED DESCRIPTION:
The overall aim of PHRASE-HF is to evaluate the use of GDMT at hospital discharge, the translation of in-hospital implementation and possible maximisation of phenotype-based GDMT into real-world routine outpatient care, HF symptoms, patient reported outcomes (PROs), clinically relevant outcomes (e.g. rehospitalisation, mortality), use of diuretics and concomitant drug classes in patients admitted for in-hospital treatment of HFrEF to sites trained within the Helios-GDMT-program. The analyses will primarily be done in a total study population, and as defined by exploratory objectives in subgroups of interest.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years at the time of signing the informed consent
* Hospitalised in a participating site and receiving full inpatient treatment (at least 24h hospital stay)
* Diagnosis of HFrEF according to the current guidelines of the European Society of Cardiology (ESC) with a left ventricular EF of ≤40% (as measured per echocardiography during the index hospital stay or within 3 months prior to index hospitalisation with available reports from imaging (ejection fraction) at the time of study inclusion)
* Treated with a maximum of 2 of the indicated drug classes (ACE-I/ARNI/ARB, BB, MRA, SGLT2i) according to guideline recommendation (GDMT) at admission.
* Signed and dated written informed consent prior to enrolment in the study
* Willing and capable to fulfil requirements listed in the ICF

Exclusion Criteria:

* Initial presentation (index hospitalisation) in cardiogenic shock or other kinds of shock
* Status post heart transplantation
* History of intolerance to one or more GDMT drug classes (ACE-I/ARNI/ARB, BB, MRA, SGLT2i) or significant side effects that led to the discontinuation of two or more substances within one drug class (except from ACE-I/ARB, e.g., if 2 different ACE inhibitors triggered cough, but sartans are tolerated, then the patient is not excluded)
* Current or planned participation in a clinical trial
* Decision by the investigator that the participant should not participate in the study if the participant is unlikely to comply with study procedures
* Pregnancy or breast-feeding

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 438 patients with reduced ejection fraction (HFrEF) admitted for in-hospital treatment with a maximum of 2 of the indicated guideline recommended drug classes (ACE-I/ARNI/ARB, BB, MRA, SGLT2i) in the current medication plan are planned to be enrolled consecutively. Recruitment will take place at 5-7 inpatient cardiology departments at Helios hospitals trained by Helios-GDMT-Program throughout Germany.
Sampling Method: Non-Probability Sample
Enrollment: 438 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients treated with HFrEF GDMT | Baseline to hospital discharge, on average 6 days after hospitalization/baseline
  Proportion of patients treated with phenotype-concordant guideline-recommended HF drug classes and the corresponding doses as noted in patients electronic medical records

SECONDARY OUTCOMES:
Number of recommended HF-drug classes | Baseline to hospital discharge, on average 6 days after hospitalization/baseline
  The HF-drug classes including the corresponding doses that are recommended in discharge letter at hospital discharge
Change of percentage in HFrEF GDMT | Baseline to 12 months
  The percentage of patients who are newly initiated on guideline-directed HFrEF medical therapy
Change of phenotype-concordant guideline-recommended HF drug classes | Hospital Discharge (on average 6 days after hospitalization/baseline) to 12 months
  The number of patients with change in phenotype-concordant guideline- recommended HF drug classes
Reasons for GDMT adjustments | Hospital Discharge (on average 6 days after hospitalization/baseline) to 12 months
  The reasons for guideline-directed medical therapy changes as noted in patients electronic medical records will be described as the number and proportion of patients who experienced adjustment in guideline-directed medical therapy according to each reasons presented
Reasons for not having guideline-recommended drug classes or doses | Hospital Discharge (on average 6 days after hospitalization/baseline) to 12 months
  The reasons for not having maximal phenotype-concordant guideline-recommended HF drug classes as noted in patients electronic medical records will be described as the number and proportion of patients who are not having maximal GDMT drug classes according to each reasons presented
Number of outpatient post-discharge visits | Hospital Discharge (on average 6 days after hospitalization/baseline) to 3 months
  The number of outpatient visits for heart failure treatment within the first three months after hospital discharge
Proportion of patients conducting post-discharge visits | Hospital Discharge (on average 6 days after hospitalization/baseline) to 3 months
  Proportion of patients conducting post-discharge visits for heart failure treatment within the first three months after hospital discharge
Absolute change from baseline in NYHA class | Measured at 6 and 12 months
  The NYHA classification is a regimen for the classification of heart failure into certain stages according to clearly defined criteria. Treatment of heart failure is usually based on the NYHA classification. Symptoms used to evaluate the stages include dyspnea, nocturia at night, cyanosis, general weakness and fatigue, angina pectoris or cold extremities, edema. NYHA-I: No limitation on resilience. Complete absence of symptoms or signs of exertion when heart disease is diagnosed; NYHA-II: Slight decrease in endurance. Freedom from discomfort during rest and with mild exertion, occurrence of symptoms with increased stress; NYHA-III: Severe limitation of resilience. Freedom from discomfort at rest, occurrence of symptoms even with mild exertion; NYHA-IV: Permanent symptoms, even during rest.
Change from Baseline in blood pressure | Baseline to 12 months
  Changes in patients blood pressure as noted in patients electronic medical records /
Change from Baseline in heart rate | Baseline to 12 months
  Changes in patients heart rate as noted in patients electronic medical records
Change from Baseline in electrolyte level | Baseline to 12 months
  Changes in patients electrolyte level as noted in patients electronic medical records
Change from Baseline in potassium level | Baseline to 12 months
  Changes in patients potassium level as noted in patients electronic medical records
Change from Baseline in estimated glomerular filtrations rate | Baseline to 12 months
  Changes in patients estimated glomerular filtration rate as noted in patients electronic medical records
Change from Baseline in serum creatinine concentration | Baseline to 12 months
  Changes in patients serum creatinine concentration as noted in patients electronic medical records
Number of rehospitalization for heart failure | Hospital Discharge (on average 6 days after hospitalization/baseline) to 12 months
  The number of patients being rehospitalized for heart failure within the observational period
Overall Survival | Baseline to 12 months
  Number of patients who died during the observational period
CV-specific survival | Baseline to 12 months
  Number of patients who died due to cardiovascular disease during observation period
Absolute change from baseline in Medication Adherence Report Scale (MARS)-5 questionnaire | Measured at 6 and 12 months
  The MARS-5 is five-item self-report adherence scale which assesses both intentional and non-intentional non-adherence. Respondents rate the frequency with which the five different medication-taking behaviours occur, scoring each item on a 1-5-point scale with higher scores indicating higher reported adherence. The MARS-5 has been shown to be reliable and valid across a variety of health conditions, including cardiovascular and pulmonary diseases. Only applicable to Prospective cohort.
Absolute change from baseline in Kansas City Cardiomyopathy Questionnaire (KCCQ) score | Measured at 6 and 12 months
  The KCCQ is a 23-item questionnaire that quantifies physical limitations, self-efficacy, social interference and quality of life. Summary scores will be examined at each assessment point during follow-up. For each of the assessment periods, descriptive statistics for the observed value, change from baseline and the 95% two-sided confidence interval for the mean change will be presented. The proportions of participants with overall health status classified as poor, fair, good, and excellent will be examined at each assessment point. Additionally, the proportions of participants who experience clinically meaningful changes in overall health status: improvement (≥5 point increase), deterioration (≥5 point decrease), and stable (<5 point increase or decrease) will be examined at each assessment point. Only applicable to Prospective cohort
Absolute change from baseline in PROMIS Global Health 10 | Measured at 6 and 12 months
  The PROMIS 10 is a validated comprehensive and accessible set of tools used to measure self-reported physical, mental and social health; including symptoms, function and general perceptions of health and wellbeing. The PROMIS 10 consists of ten items that measure physical health, physical functioning, general mental health, emotional distress, satisfaction with social activities and relationships, ability to carry out usual social activities and roles, pain, fatigue and overall quality of life.
Absolute change from baseline in the Nine-Item Patient Health Questionnaire (PHQ-9) | Measured at 6 and 12 months
  HF is associated with depressive disorders and manifest depressions. The PHQ-9 that capture depressed mood and anhedonia has been validated as an ultra-brief screening tool with some evidence of responsiveness. The PHQ-9 score is obtained by adding the score for each question (total points). A PHQ-9 score ranges from 0-27, to determine whether they meet criteria for a depressive disorder.
Number of diuretics changes | Baseline to 12 months
  The number of patients who experience a switch in their diuretic medication drug class as noted in patients electronic medical record
Number of concomitant medication changes | Baseline to 12 months
  The number of patients who experience a switch in their concomitant medication drug class as noted in patients electronic medical record

CONTACTS AND LOCATIONS:
Locations (6):
- Germany (6):
  - Research Site, Berlin
  - Research Site, Erfurt
  - Research Site, Gifhorn
  - Research Site, Leipzig
  - Research Site, Schwerin
  - Research Site, Wuppertal

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm/ST/Submission/Disclosure Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm/ST/Submission/Disclosure
Access Criteria: When a request has been approved, AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm/ST/Submission/Disclosure
URL: https://vivli.org/